CLINICAL TRIAL: NCT05367791
Title: Improving Postural Control Through Innovative Stimulation of the Proprioceptive System
Acronym: IMPULSES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21CH160; 2021-A02416-35 (Other: ANSM)
Record Dates: First submitted 2022-05-02; First posted 2022-05-10 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Sensorimotor Disorder
Keywords: Postural exercise; Localized vibration; Somatosensory electrical stimulation; Altered posture; Walking control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- POSTUR (Other): Postural training only.
  Interventions: Other: POSTUR
- POSTUR + LV (localized vibration) (Other): Postural training combined with localized vibration
  Interventions: Other: POSTUR; Other: Localised Vibration
- POSTUR+SES (somatosensory electrical stimulation) (Other): Postural training combined with somatosensory electrical stimulation
  Interventions: Other: POSTUR; Other: Somatosensory Electrical Stimulation
- POSTUR+LV-SES (Other): Postural training combined with somatosensory electrical stimulation and localized vibration
  Interventions: Other: POSTUR; Other: Localised Vibration; Other: Somatosensory Electrical Stimulation

INTERVENTIONS:
Other: POSTUR — Training sessions without any stimulation
Other: Localised Vibration — Training sessions with localized vibration
  Arms: POSTUR + LV (localized vibration); POSTUR+LV-SES
Other: Somatosensory Electrical Stimulation — Training sessions with somatosensory electrical stimulation
  Arms: POSTUR+LV-SES; POSTUR+SES (somatosensory electrical stimulation)

SUMMARY:
Every movement humans make in everyday life is based on a continuous integration of sensory information. A good interaction between sensory processes and motor control, called sensorimotor integration, is necessary for the efficiency of movements. Sensorimotor integration in the context of posture and walking is based on proprioception. Proprioception is the conscious and unconscious perception of the spatial and mechanical state of the musculoskeletal system. Proprioceptive information transmitted through the neuromuscular spindles in particular is suggested to play a role in motor rehabilitation.

DETAILED DESCRIPTION:
This is particularly important when considering populations with impaired proprioception resulting in impaired posture and gait control. This is particularly the case for older adults and children with cerebral palsy (CP). Nevertheless, drastic differences exist between the two populations in the nature of these alterations: stable (children with CP) vs. progressive (older adults); brain lesion/upper motor neuron (children with CP) vs. processing deficits and peripheral sensory degradation (older adults); growing (children with CP) vs. fully developed individuals (older adults). However, both populations can improve their postural control with postural exercise programmes. In humans, the proprioceptive system can also be stimulated non-invasively by mechanical vibrations applied to tendons or muscles (localised vibration; LV), or by electrical stimulation of peripheral nerves (somatosensory electrical stimulation; SES). As a result, chronically applied SES can improve sensorimotor function in healthy adults and some clinical cohorts. Similarly, a 6-week weight-bearing and weight-shifting training programme combined with LV has been reported to provide improved benefits in postural control, again in stroke patients.The greater improvement in motor function when LV or SES is added to active muscles may reflect an adjuvant effect: the sensory signal from LV or SES stimulation is integrated with the sensory signals from the task being performed, thus acting as an associative conditioning of the proprioceptive system, and leading to improved sensorimotor integration. The present project aims to study the effectiveness of a short-term intervention combining postural exercises with LV, SES, or the combination of both.

In particular, this study will focus on the effects of these interventions on proprioception, postural control and walking in children with CP and older adults.Confirmation of hypotheses will open up new avenues for rehabilitation therapies and preventive interventions, and may be extended to other purposes and clinical populations.

ELIGIBILITY:
Inclusion Criteria:

Older Adults:

* Affiliated or beneficiaries of a social security plan
* Who have freely given their written consent after having been informed of the purpose, the procedure and the potential risks involved

Children with Cerebral Palsy:

* Children between the ages of 7 and 18 years, diagnosed with Spastic Cerebral Palsy, presenting with a clinical picture of infantile cerebral hemiplegia or diplegia.
* Children able to understand and follow the simple instructions of the examination
* Children walking GMFCS (Gross Motor Functional Classification system) I to II.
* Children with at least one parent and the child having given and signed the consent agreement
* Children who are members or beneficiaries of a social security system

Exclusion Criteria:

Older adults:

* Pathology or surgery resulting in a locomotor disorder, within 6 months prior to the study,
* Chronic neurological, motor or psychological pathologies
* Use of neuro-active substances likely to alter cortico-spinal excitability (hypnotics, anti-epileptics, psychotropic drugs, muscle relaxants) during the study.
* Contraindication to transcranial magnetic stimulation:

  * Cardiac or respiratory insufficiency.
  * Wearing a cardiac pace maker.
  * Wearing a heart valve and severe cardiovascular diseases.
  * Presence of prosthetic material or ferromagnetic foreign bodies in the head.
  * Presence of cochlear implants or ocular prosthetic material.
  * History of neurosurgical procedures.
  * Neurological diseases that may affect brain structures and cognitive abilities (e.g., intracranial tumor, multiple sclerosis, history of stroke or head injury).
* Participation at the same time in another interventional trial or having participated in a such a study within 30 days prior to this study.
* Obesity (body mass index ≥ 30.0 kg/m²)

Children with cerebral palsy:

* Children with concomitant muscle disease (e.g., myopathy...).
* Children who have received a baclofen injection in the 6 months preceding the evaluation.
* Children who have undergone neuro-orthopedic surgery on the lower limbs within the last 6 months
* Children who have received a botulinum toxin injection within the last 6 months
* Children participating in therapeutic programs other than their usual physical therapy sessions.

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-07-22 (Actual)

PRIMARY OUTCOMES:
Evaluation of body balance with the Berg Balance Scale (BBS) | Change from Week 8 to Week 16
  Variation of postural control

SECONDARY OUTCOMES:
Evaluation of body balance with the Berg Balance Scale (BBS) | Change from Week 1 to Week 22
  Variation of postural control
Evaluation of the displacement of the center of pressure with force platform in centimeter | Change from Week 1 to Week 22
  Variation of postural control
Displacement of the centrer of pressure with application of localized vibration in centimeter | Change from Week 1 to Week 22
  Proprioceptive contribution to postural control
Measure of the angular position error in degrees | Change from Week 1 to Week 22
  Variation of the position direction
Coefficient of variation muscle force control in percent | Change from Week 1 to Week 22
  Muscle force control measurement
Measure 6-minute walk test (6MWT) in meters | Change from Week 1 to Week 22
  Walking ability evaluation
Measure Timed Up & Go Test (TUG) in seconds | Change from Week 1 to Week 22
  Walking ability evaluation
Measure 10 meter walk test (10MWT) in seconds | Change from Week 1 to Week 22
  Walking ability evaluation
Quantifying corticospinal excitability with motor evoked potentials in milliVolt | Change from Week 1 to Week 22
  Underlying neural adaptations evaluation in older adults only
Quantifying spinal excitability with H-reflex in milliVolt | Change from Week 1 to Week 22
  Underlying neural adaptations evaluation in older adults only

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Feasson, PHD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- Centre Hospitalier de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No